CLINICAL TRIAL: NCT05723783
Title: The Prognostic Value of CT-guided Sarcopenia for Surgical Outcomes in Patients Submitted to Esophagetomy and Total Gastrectomy Due to Neoplasia
Brief Title: Prognostic Value of CT-guided Sarcopenia for Surgical Outcomes in Esophagetomy and Total Gastrectomy Due to Neoplasia
Status: Completed | Type: Observational
Sponsor: Barretos Cancer Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: BarretosCH
Record Dates: First submitted 2018-08-21; First posted 2023-02-13 (Actual); Last update posted 2023-02-13 (Actual); Status verified 2023-02

CONDITIONS: Sarcopenia; Malnutrition; Gastrostomy; Esophagostomy Complication; Computed Tomography
Keywords: sarcopenia; cancer; gastrectomy; esophagectomy; computed tomography; morbidity; mortality; malnutrition
MeSH Terms: conditions — Sarcopenia; Malnutrition; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
The purpose of this study is to assess the degree of sarcopenia by CT and to analyze its association with morbidity and mortality after esophagectomy and / or total gastrectomy. It is also intended to analyze the association between the degree of the CT-guided sarcopenia and the nutritional status of the patients evaluated by clinical parameters, both preoperative and postoperative. Besides that, to verify the association between the degree of sarcopenia and body fat rate.

DETAILED DESCRIPTION:
Background: Malnutrition is highly prevalent in patients with esophageal and / or stomach cancer, and is often followed by sarcopenia (loss of muscle mass and strength). Both syndromes influence negatively on prognosis of oncological patients, by increasing hospitalization time, number of complications and hospital expenses. Therefore, it is extremely important to identify patients at nutritional risk. This nutritional assessment can be done through clinical and laboratory tests, as well as can be inferred through computed tomography (CT) imaging.

Hypothesis: To evaluate the relationship between the rate of CT-guided sarcopenia and the surgery outcomes of patients undergoing esophagectomy and / or total gastrectomy due to neoplasia.

Methods: Prospective non-randomized study evaluating the nutritional status and morbidity and mortality of patients. The cases will be conducted according to a pre-established protocol and the sample, for convenience, will be 80 patients. Demographic data and information on diagnosis, treatment and post-surgical data will be collected, as well as anthropometric evaluation. In addition, biochemical data such as hemoglobin, transferrin and serum albumin values will be assessed to classify the patient's nutritional status. The CT images will be analyzed in order to evaluate the degree of sarcopenia and body fat rate, using the distal sections of the third lumbar vertebra. In order to evaluate skeletal muscle mass, the areas of interest will be ones between -30 and +110 hounsfield units (HU) and for the analysis of visceral fat area analysis, pixels with densities between -190 to -30 HU will be used. Both results will be converted to cm2 and analyzed through pre-set cutoff values.

Statistical analysis: Descriptive analyzes will be performed using Fisher's exact tests, for proportions; Wilkcoxon rank-sum test for analyzes of continuous and non-parametric variables. Univariate analyzes will be performed to compare the variables of interest of the study, with the other variables. All tests will have a 5% significance level.

ELIGIBILITY:
Inclusion Criteria:

* elective esophagectomy and / or total gastrectomy due to neoplasia,
* received oral or enteral diet in less than 48 hours postoperatively. For those who started with an enteral catheter, will be included in the study those with oral feedback up to 7 days.

Exclusion Criteria:

* Need for colonic transposition instead of gastric tube for reconstruction;
* Presence of any adverse events related to the anesthetic act or not related to the surgical act.

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients of Barretos Cancer Hospital with primary esophageal or gastric cancer, undergoing surgical treatment on this institution.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2017-01-20 (Actual); Primary Completion 2018-12-20 (Actual); Study Completion 2019-01-20 (Actual)

PRIMARY OUTCOMES:
Degree of sarcopenia | Preoperative - around 30 days before surgery
  To assess skeletal muscle mass, areas of interest were considered those between -29 to +150 Hounsfield Units (HU), and converted to cm². The final value obtained was the skeletal muscle mass index (cm²/m²) (MMI), calculated by dividing the value obtained by height (m) squared and classified according to the cut-off points established.
Morbidity and mortality | Postoperative - 30 days after surgery
  Number of complications according to the scale of clavien-dindo after esophagectomy and / or total gastrectomy

SECONDARY OUTCOMES:
Nutritional status | Preoperative, days 30, 60 and 90 postoperative
  Analyze the nutritional status of the patients evaluated by clinical parameters (weight in kilograms and height in meters will be combined to report Body Mass Index in kg/m²).
Evolution of serum dosage of hemoglobin albumin and transferrin | Preoperative, days 30, 60 and 90 postoperative
  Analyze biochemical parameters: serum levels of albumina (g/dL), transferrina (mg/dL) and hemoglobina (g/dL).
Total, visceral and subcutaneous fat area by CT | preoperative around 30 days before surgery
  Total fat area (TFA) and visceral fat area (VFA) were evaluated by measuring pixels with densities between -190 to -30 Hounsfield Units in cm². Subcutaneous fat area was calculated from AGT subtraction of AGT.

CONTACTS AND LOCATIONS:
Overall Officials: Raphael LC Araújo, PHD, Principal Investigator — Cancer Hospital Barretos
Locations (1):
- Barretos Cancer Hospital, Barretos, São Paulo, Brazil